CLINICAL TRIAL: NCT07297927
Title: Prospective Study on ICG Lymphoscintigraphy Changes Before and After Radiotherapy in Breast Cancer Patients
Acronym: ICG_prepostRT
Status: Recruiting | Type: Observational
Sponsor: Inah Kim (Other)
Responsible Party: Sponsor-Investigator, Inah Kim, Clinical Assistant Professor, Dongtan Sacred Heart Hospital
Organization: Dongtan Sacred Heart Hospital (Other)
Other Study IDs: 2025-10-008
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Breast Neoplasms; Lymphedema Due to Radiation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn how the lymphatic system changes before and after radiotherapy in female patients with breast cancer. The study aims to understand early lymphatic changes that may lead to breast-cancer-related lymphedema (BCRL) and to help identify patients who might benefit from early preventive rehabilitation.

The main questions it aims to answer are:

How does lymphatic flow and vessel function change after radiotherapy, as measured by indocyanine green (ICG) lymphography?

Can early imaging changes on ICG lymphography predict later swelling or lymphedema symptoms in the arm?

There is no comparison or treatment group, since all participants will receive radiotherapy as part of their standard breast cancer care.

Participants will:

Undergo ICG lymphography before radiotherapy and again within 4-6 weeks after completing radiotherapy

Receive a small injection of ICG dye under the skin and have near-infrared imaging to visualize lymphatic flow

Complete follow-up assessments (for some participants) at 3, 6, or 12 months to monitor long-term lymphatic changes

Continue their usual standard medical and rehabilitation care throughout the study

This study will include 40 female participants, aged 18 years or older, who have been diagnosed with stage I-III breast cancer and are scheduled for postoperative radiotherapy. Participants with a history of lymphedema, prior radiotherapy, severe organ disease, or known ICG/iodine allergy will not be included.

The information collected will include imaging findings from ICG lymphography, arm circumference and volume measurements, and patient-reported outcomes on arm discomfort or swelling. These data will help researchers identify early imaging biomarkers of radiation-induced lymphatic dysfunction.

The study does not involve any experimental treatment or random assignment. All procedures are routine diagnostic or rehabilitation methods that are already approved for clinical use. The ICG test uses a very small amount of dye and is considered safe, with allergic reactions being rare.

The findings of this study may provide new insights into how radiotherapy affects the lymphatic system and may contribute to developing personalized strategies to prevent or minimize lymphedema after breast cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female, ≥18 years old Pathologically confirmed stage I-III breast cancer Scheduled to receive postoperative radiotherapy (RT)

Exclusion Criteria:

* Previous or current lymphedema Prior radiotherapy to the ipsilateral breast or axilla History of neoadjuvant chemotherapy Severe systemic diseases (heart, renal, hepatic failure) Active infection Pregnancy or lactation Allergy to indocyanine green (ICG) or iodine-based contrast agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female breast cancer survivors (stage I-III) scheduled for adjuvant radiotherapy after surgery. Participants are recruited consecutively from the Department of Rehabilitation Medicine, Radiation Oncology and General Surgery at Hallym University Dongtan Sacred Heart Hospital. The study population represents patients at risk for radiation-induced lymphatic dysfunction or breast-cancer-related lymphedema.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2028-10-18 (Estimated)

PRIMARY OUTCOMES:
Change in Lymphatic Function Before and After Radiotherapy Measured by ICG Lymphography | Baseline (before radiotherapy), 4-6 weeks after completion of radiotherapy, and optionally at 3, 6, and 12 months after RT completion if follow-up imaging is performed.
  Quantitative and qualitative changes in lymphatic function assessed by indocyanine green (ICG) lymphography before and after radiotherapy (RT). Parameters include uptake pattern, lymphatic contractility, fluorescence intensity, and dermal backflow pattern. These measures reflect radiation-induced lymphatic dysfunction and may serve as early imaging biomarkers for breast-cancer-related lymphedema (BCRL).

SECONDARY OUTCOMES:
Change in Arm Circumference and Limb Volume After Radiotherapy | Baseline (before radiotherapy), 4-6 weeks, and optionally at 3, 6, and 12 months after RT completion
  Change in arm circumference and estimated limb volume (using the truncated cone formula) before and after radiotherapy (RT), compared with baseline measurements. These measurements will be used to determine whether early lymphatic imaging changes are correlated with the development or progression of breast-cancer-related lymphedema (BCRL).

CONTACTS AND LOCATIONS:
Locations (1):
- Dongtan Sacred Heart Hospital, Hwaseong-si, Gyeonggido, South Korea

IPD SHARING:
Plan to Share IPD: No